CLINICAL TRIAL: NCT05215652
Title: Adherence Monitoring Package to Identify Non-adherence in Ambulatory Hypertensive Patients
Brief Title: Adherence Monitoring in Ambulatory Hypertensive Patients
Acronym: AMoPac-HYP
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: 2021-02392
Record Dates: First submitted 2022-01-18; First posted 2022-01-31 (Actual); Last update posted 2023-04-27 (Actual); Status verified 2023-04

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: adherence monitoring package (AMoPac) — AMoPac is a tool that consists of
  * an electronic monitoring device,
  * data management and data analysis,
  * feedback on patient's performance,
  * clinical-pharmaceutical evaluation of medication adherence,
  * transmission of an adherence report.

SUMMARY:
Hypertension is a major risk factor for stroke, ischaemic heart disease, and kidney disease. One major cause for uncontrolled blood pressure in spite of prescribed pharmacotherapy was found to be non-adherence including erratic use of prescribed medication.

General practitioners (GP) face limitations when a guideline-conform therapy fails. A new tool to measure and assess medication adherence could be useful to identify patients who are not using medicine as prescribed. This provides new opportunities for patient-specific recommendations and adjustments of treatment.

Our aim is to assess the usefulness of the adherence package AMoPac to identify non-adherence in hypertensive patients nonresponding to treatment in daily practice.

DETAILED DESCRIPTION:
Patients with hypertension are usually asymptomatic and do not feel an immediate benefit when taking their medication. This can result in early treatment interruption, omitted doses or drug holidays. Especially when side effects occur, which is often reported for diuretics and ACE inhibitors, patients tend to take their medicines less regularly or even to omit them. Furthermore, it is known that adherence decreases with the increased number of daily medicines. Patients with polypharmacy are thus particularly affected by non-adherence, that is almost inevitable in hypertensive treatment using dual, triple or quadruple therapy. Erratic use of prescribed medication including non-adherence is a major cause for uncontrolled blood pressure. However, practical and reliable methods are missing to screen patients for non-adherence.

The investigators have developed the adherence monitoring package (AMoPac) to help identifying non-adherence in ambulatory hypertensive patients. AMoPac is a tool that consists of an electronic monitoring device (Time4Med™ or smart phone application), data management and data analysis, feedback on patient's performance and clinical-pharmaceutical evaluation of medication adherence. The purpose is to transmit a patient-specific adherence report (including adherence recommendations) to the the GP.

This study is a prospective, observational study. GPs will recruit hypertensive patients during their routine visits. Patients will monitor daily medication intake at home for 4 weeks. A pharmacist will visit the patient at home to download the adherence data and to give feedback. The patient will then visit the GP who will have already received the adherence report and will have the opportunity to intervene, for example by adapting the patient's treatment or their medication use behavior. The 4-weeks cycle of adherence monitoring can be repeated if needed.

The investigators expect that AMoPac is useful for GPs to identify non-adherence in hypertensive patients nonresponding to treatment.

ELIGIBILITY:
Inclusion Criteria:

Patients with the following inclusion criteria will be recruited:

* is ≥18 years old;
* is diagnosed with arterial hypertension;
* is prescribed at least 1 antihypertensive medication;
* self-administers medication;
* is suspected of a deviant medication intake behavior (non-adherence) e.g., because of insufficiently controlled blood pressure in spite of prescribed pharmacotherapy (nonresponding);
* accepts to use of an electronic monitoring device during the study period (either the Time4Med™ device or the monitoring app busybee™);
* signs the informed consent form;
* understands and speaks German.

Patients who are using a pillbox, an app or reminders for medication management will not be excluded.

Exclusion Criteria:

Patients who are, in the opinion of the GP, unlikely to comply with the study schedule or are unsuitable for any other reason will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: hypertensive patients nonresponding to pharmacotherapy
Sampling Method: Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2022-02-15 (Actual); Primary Completion 2023-04-17 (Actual); Study Completion 2023-04-17 (Actual)

PRIMARY OUTCOMES:
Usefulness of the adherence package AMoPac | through study completion, 1 year
  The primary objective is to assess the usefulness of the adherence package AMoPac to identify non-adherence in hypertensive patients nonresponding to treatment in daily practice. It is defined as ≥75% of participating GPs who rate that the AMoPac is useful to identify hypertensive patients nonresponding to treatment as non-adherent.

SECONDARY OUTCOMES:
errors in medication use | one month
  the types of critical errors in medication use made by hypertensive patients
treatment adaptions | one month
  the impact of AMoPac on clinical decision-making (questionnaire)
Adherence counselling | one month
  the impact of AMoPac on medication intake behaviour counselling (questionnaire)
Medication adherence | one month
  the level of patient medication adherence (metrics: taking and timing adherence, correct dosing days)
Blood pressure | one month
  the level of patient blood pressure control, measured at GP office at study entry and end-of-study visit
Patient satisfaction | one month
  patient satisfaction with the electronic adherence monitoring (questionnaire)

CONTACTS AND LOCATIONS:
Locations (1):
- Praxis Hammer, Basel, Switzerland